CLINICAL TRIAL: NCT00947908
Title: Regulation of Blood Dendritic Cells During Immune Therapy for Hymenoptera Venom Allergy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Rostock (Other)
Responsible Party: PD Dr. Marek Lommatzsch, University of Rostock
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LO-0004
Record Dates: First submitted 2009-07-27; First posted 2009-07-28 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2009-07

CONDITIONS: Hymenoptera Venom Allergy
Keywords: Hymenoptera venom allergy; Dendritic cells (DC)
MeSH Terms: interventions — Arthropod Venoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Patients are treated with hymenoptera (bee or wasp) venom using subcutaneous injections. The initiation of immune therapy consists of a 52-hour-period in which patients are treated with increasing doses of hymenoptera venom. Afterwards, patients are treated with monthly subcutaneous injections with a fixed dose of hymenoptera venom. Blood will be collected directly before and 1 hour after initiation of immune therapy and after 12 months of immune therapy (directly before the next subcutaneous injection of hymenoptera venom).
  Interventions: Biological: Hymenoptera venom

INTERVENTIONS:
Biological: Hymenoptera venom — Patients are treated with hymenoptera (bee or wasp) venom using subcutaneous injections. The initiation of immune therapy consists of a 52-hour-period in which patients are treated with increasing doses of hymenoptera venom. Afterwards, patients are treated with monthly subcutaneous injections with a fixed dose of hymenoptera venom. Blood will be collected directly before and 1 hour after initiation of immune therapy and after 12 months of immune therapy (directly before the next subcutaneous injection of hymenoptera venom).

SUMMARY:
Dendritic cells (DC) play a key role in the pathogenesis of allergic diseases. The regulation of blood dendritic cells in patients with hymenoptera venom allergy before and during immune therapy is unknown.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed hymenoptera venom allergy
* No previous treatments for hymenoptera venom allergy

Exclusion Criteria:

* Treatment with immunosuppressive agents
* Any malignant disease
* Infections within 1 week prior to the initiation of the treatment

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Number of myeloid DC and plasmacytoid DC in peripheral blood | Directly before, 1 hour after, and 12 months after initiation of immune therapy

SECONDARY OUTCOMES:
Surface molecule expression on myeloid DC and plasmacytoid DC | Directly before, 1 hour after, and 12 months after initiation of immune therapy

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rostock, Rostock, Mecklenburg-Vorpommern, Germany

REFERENCES:
- [Background] Bratke K, Lommatzsch M, Julius P, Kuepper M, Kleine HD, Luttmann W, Christian Virchow J. Dendritic cell subsets in human bronchoalveolar lavage fluid after segmental allergen challenge. Thorax. 2007 Feb;62(2):168-75. doi: 10.1136/thx.2006.067793. Epub 2006 Aug 23. PMID 16928719
- [Derived] Dreschler K, Bratke K, Petermann S, Bier A, Thamm P, Kuepper M, Virchow JC, Lommatzsch M. Impact of immunotherapy on blood dendritic cells in patients with Hymenoptera venom allergy. J Allergy Clin Immunol. 2011 Feb;127(2):487-494.e1-3. doi: 10.1016/j.jaci.2010.12.003. PMID 21281873